CLINICAL TRIAL: NCT06219941
Title: A Phase II, Open-label, Multi-centre Study to Evaluate Safety, Tolerability, Efficacy, PK, and Immunogenicity of AZD0901 as Monotherapy and in Combination With Anti-cancer Agents in Participants With Advanced Solid Tumours Expressing Claudin 18.2 (CLARITY-PanTumour01)
Brief Title: AZD0901 in Participants With Advanced Solid Tumours Expressing Claudin18.2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9800C00001
Record Dates: First submitted 2023-11-21; First posted 2024-01-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer; Biliary Tract Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: Gastric cancer; Gastroesophageal junction cancer; Pancreatic Ductal adenocarcinoma; Biliary Tract Cancer; Phase II; Claudin 18.2; AZD0901
MeSH Terms: conditions — Stomach Neoplasms; Biliary Tract Neoplasms | interventions — Fluorouracil; Leucovorin; Irinotecan; irinotecan sucrosofate; Gemcitabine

STUDY DESIGN:
Intervention Model Description: This study is an open-label, multi-centre study of AZD0901 administered via IV, either as monotherapy or in combination with other anti-cancer agents in participants with advanced solid malignancies expressing CLDN18.2. The substudy design allows for a targeted approach to the different tumour types as monotherapy or in combination with other anti-cancer agents. These substudies include:
  Substudy 1: AZD0901 monotherapy in gastric and gastric esophageal junction cancer patients Substudy 2: AZD0901 in combination with anti-cancer agents in pancreatic cancer patients.
  Substudy 3: AZD0901 monotherapy in biliary Tract Cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sub Study 1 - AZD0901 MONOTHERAPY (Experimental): Sub Study 1 will investigate AZD0901 monotherapy in order to evaluate the safety, tolerability, and efficacy of AZD0901.
  Interventions: Drug: AZD0901
- Sub Study 2 - AZD0901 IN COMBINATION WITH ANTI-CANCER AGENTS IN PANCREATIC DUCTAL ADENOCARCINOMA (Experimental): Substudy 2 will investigate the safety and efficacy of AZD0901 as first line systemic treatment used in combination with different chemotherapy agents
  Interventions: Drug: AZD0901; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: l-leucovorin; Drug: Irinotecan; Drug: Nanoliposomal Irinotecan; Drug: Gemcitabine
- Sub Study 3: AZD0901 MONOTHERAPY IN BILIARY TRACT CANCER (Experimental): Substudy 3 Further evaluate the preliminary anti-tumour activity of AZD0901 monotherapy by assessment of DRR.
  Interventions: Drug: AZD0901

INTERVENTIONS:
Drug: AZD0901 — Antibody-drug conjugate/Biologic
  Other Names: CMG901
Drug: 5-Fluorouracil — Chemotherapy agents
  Other Names: 5-FU
  Arms: Sub Study 2 - AZD0901 IN COMBINATION WITH ANTI-CANCER AGENTS IN PANCREATIC DUCTAL ADENOCARCINOMA
Drug: Leucovorin — Chemotherapy agents
  Other Names: LV
  Arms: Sub Study 2 - AZD0901 IN COMBINATION WITH ANTI-CANCER AGENTS IN PANCREATIC DUCTAL ADENOCARCINOMA
Drug: l-leucovorin — Chemotherapy agents
  Other Names: I-LV
  Arms: Sub Study 2 - AZD0901 IN COMBINATION WITH ANTI-CANCER AGENTS IN PANCREATIC DUCTAL ADENOCARCINOMA
Drug: Irinotecan — Chemotherapy agents
  Other Names: Camptosar
  Arms: Sub Study 2 - AZD0901 IN COMBINATION WITH ANTI-CANCER AGENTS IN PANCREATIC DUCTAL ADENOCARCINOMA
Drug: Nanoliposomal Irinotecan — Chemotherapy agents
  Other Names: ONIVYDE
  Arms: Sub Study 2 - AZD0901 IN COMBINATION WITH ANTI-CANCER AGENTS IN PANCREATIC DUCTAL ADENOCARCINOMA
Drug: Gemcitabine — Chemotherapy agents
  Other Names: Gemzar
  Arms: Sub Study 2 - AZD0901 IN COMBINATION WITH ANTI-CANCER AGENTS IN PANCREATIC DUCTAL ADENOCARCINOMA

SUMMARY:
The purpose of this study is to assess the safety, tolerability, efficacy, pharmacokinetics (PK), and immunogenicity of AZD0901 as monotherapy and in combination with anti-cancer agents in participants with locally advanced unresectable or metastatic solid tumours expressing CLDN18.2.

DETAILED DESCRIPTION:
This open-label, multi-centre study consists of individual sub studies, each evaluating the safety and tolerability of AZD0901.

Sub study 1 will investigate the safety, tolerability, and anti-tumour activity of AZD0901 monotherapy in participants with advanced or metastatic gastric esophageal cancer expressing CLDN18.2. Participants will receive AZD0901 monotherapy via intravenous (IV) infusion and will be randomised in to one of 2 arms.

Sub study 2 will consist of two parts, a safety run-in and a dose expansion part to investigate the safety and efficacy of AZD0901 in combination with different chemotherapy agents in participants with pancreatic cancer. Substudy 3 will investigate the safety, tolerability, and anti-tumour activity of AZD0901 monotherapy in participants with advanced or metastatic Biliary tract cancer.

ELIGIBILITY:
The list below is a summarised eligibility criteria for the study - refer to the study protocol for full criteria.

Master Inclusion Criteria applicable to all sub studies:

* Participant must be ≥ 18 years or the legal age of consent at the time of signing the ICF.
* Participants who are CLDN18.2 positive.
* Must have at least one measurable lesion according to RECIST v1.1.
* ECOG performance status of 0 to 1 with no deterioration over the previous 2 weeks prior first day of dosing.
* Predicted life expectancy of ≥ 12 weeks.
* Adequate organ and bone marrow function as defined by protocol.
* Body weight > 35 kg.
* Participants are willing to comply with contraception requirements.

Sub study 1 Specific Inclusion criteria:

* Histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction.
* Advanced or metastatic GC/GEJC.
* Maximum 2 prior lines of systemic treatment for unresectable or metastatic disease.

Sub study 2 Specific Inclusion criteria:

* Participants diagnosed with histologically confirmed metastatic or advanced PDAC.
* Availability of an archival sample or a fresh tumour biopsy taken at screening.
* No prior treatments for unresectable or metastatic disease. Prior neoadjuvant/adjuvant chemotherapy is permitted as long as participants progressed ≥ 6 months (183 days) from the last dose.

Sub study 3 Specific Inclusion criteria

* Histologically confirmed, unresectable advanced, or metastatic adenocarcinoma of biliary tract, including cholangiocarcinoma (intrahepatic or extrahepatic) and gallbladder carcinoma (NOTE: Ampullary cancers are not eligible).
* Documented radiographic or clinical disease progression on or after at least one prior regimen and maximum 2 prior lines of systemic treatment for unresectable or metastatic disease.

Master Exclusion Criteria applicable to all sub studies:

* Unstable or active peptic ulcer disease or digestive tract bleeding including but not limited to clinically significant bleeding in the setting of prior CLDN18.2 directed therapy.
* Participants with clinically significant ascites that require drainage.
* A history of drug-induced non-infectious ILD/pneumonitis.
* Central nervous system metastases or CNS pathology.
* Peripheral neuropathy, sensory, or motor ≥ Grade 2 at screening.
* History of another primary malignancy.
* Prior exposure to any MMAE-based ADC.
* Prior exposure to any CLDN18.2 targeted agents except anti-CLDN18.2 monoclonal antibody.

Sub study 1 Specific Exclusion criteria:

* Participants with HER2-positive (3+ by IHC, or 2+ by IHC, and positive by ISH) or indeterminate GC/GEJC unless they have failed/not tolerated/or are not eligible for standard anti-HER2 therapy, where available.
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events.
* The use of concomitant medications known to prolong the QT/QTc interval.

Sub study 2 Specific Exclusion criteria:

* Known DPD enzyme deficiency based on local testing where testing is SoC.
* Use of strong inhibitor or inducer of UGT1A1.
* Use of strong inhibitors or inducers of CYP3A4.
* Known homozygous for the UGT1A1*28 allele based on local testing where testing is SoC.

Sub study 3 Specific Exclusion criteria

• Clinically significant biliary obstruction that has not resolved before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs), serious AEs (SAEs). Changes from baseline in clinical laboratory parameters, vital signs, ECGs and physical examination. Rate of AEs leading to discontinuation of AZD0901, Occurrence of DLTs. | 30 days post treatment completion. AE Follow Up for 90 days post AZD0901 discontinuation.
  To investigate the safety and tolerability, of AZD0901 monotherapy or in combination with anti-cancer agents in particpants with advanced or metastatic solid tumours expressing CLDN18.2.
Objective Response Rate (ORR). | From date of first dose of AZD0901 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years).
  Proportion of participants with a confirmed Complete Response (CR) or Partial Response (PR) as determined by the Investigator at local site as per RECIST v1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of first dose/randomisation until the date of death due to any cause (approximately 2 years).
  The analysis will include all dosed/randomised participants as assigned/randomised. All deaths will be included, regardless of whether the participant withdraws from therapy or receives another anticancer therapy.
Progression Free Survival (PFS) | From date of first dose/randomisation until disease progression or death in the absence of progression (approximately 2 years).
  Progression-free survival is defined as the time date of randomisation or enrollment until progression per RECIST v1.1 as assessed by the Investigator at local site, or death due to any cause, regardless of whether the participant withdraws from randomized therapy, receives another anti-cancer therapy or clinically progresses prior to RECIST v1.1 progression.
Duration of Response (DoR) | From the date of first documented confirmed response until date of documented progression (approximately 2 years).
  The time from the date of first documented confirmed response until date of first documented progression per RECIST v1.1 or death due to any cause.
Disease control rate (DCR) | Up to 11 weeks post date of first dose/randomisation
  The percentage of participants who have a confirmed CR or PR or who have SD per RECIST v1.1 as assessed by the Investigator at local site and derived from the raw tumour data up to 11 weeks after date of first dose/randomisation.
Percentage change in tumor size | From start through to study completion.
  The best percentage change from baseline in tumor size is the largest decrease (or smallest increase) from baseline for a participant, using RECIST v1.1 assessments.
Serum concentration of AZD0901 (total ADC), total antibody (conjugated and unconjugated) and total unconjugated MMAE | From date of first dose of AZD0901 up until 90 days post AZD0901 discontinuation.
  To characterise the PK of AZD0901 monotherapy or in combination with anti cancer agents in participants with advanced or metastatic solid tumours expressing CLDN18.2.
Serum PK parameters of AZD0901, total antibody (conjugated and unconjugated) and MMAE including but not limited to AUC, Cmax, tmax, clearance and half-life, as data allow. | From date of first dose of AZD0901 up until 90 days post AZD0901 discontinuation.
  To characterise the PK of AZD0901 monotherapy or in combination with anti cancer agents in participants with advanced or metastatic solid tumours expressing CLDN18.2.
Clinical activity by baseline and/or on-treatment tissue-based biomarkers including, but not limited to, gene expression, mutation profiles, DNA damage, protein expression, immune response and/or mechanisms of resistance. | From date of first dose of AZD0901 up to 7 weeks.
  To investigate baseline and/or on-treatment tissue-based RNA, DNA, and/or proteins, and association with clinical activity of AZD0901 (substudy 1).
ADA status will be determined along with prevalence and incidence of anti-drug antibodies to AZD0901, and titer established. | From date of first dose of AZD0901 up until 90 days post AZD0901 discontinuation.
  To determine the immunogenicity of AZD0901 monotherapy or in combination with anti-cancer agents in participants with advanced or metastatic solid tumours expressing CLDN18.2.

CONTACTS AND LOCATIONS:
Locations (46):
- United States (7):
  - Research Site, Orange, California
  - Research Site, Palo Alto, California
  - Research Site, Santa Rosa, California
  - Research Site, Louisville, Kentucky
  - Research Site, Commack, New York
  - Research Site, Providence, Rhode Island
  - Research Site, Houston, Texas
- Australia (3):
  - Research Site, Melbourne
  - Research Site, Murdoch
  - Research Site, Randwick
- Canada (4):
  - Research Site, Kingston, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec
- China (2):
  - Research Site, Changsha
  - Research Site, Chengdu
- Research Site, Tbilisi, Georgia
- Japan (6):
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Nagoya
  - Research Site, Osakasayama-shi
- Malaysia (5):
  - Research Site, George Town
  - Research Site, Johor Bahru
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Kuching
- Research Site, Chisinau, Moldova
- Poland (2):
  - Research Site, Krakow
  - Research Site, Warsaw
- Singapore (2):
  - Research Site, Bukit Merah
  - Research Site, Singapore
- South Korea (2):
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (4):
  - Research Site, Glasgow
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home